CLINICAL TRIAL: NCT01346215
Title: Study of Clinical Non-inferiority of Actparin® (Laboratorio Bergamo) Compared to Heparin Sodium (APP Pharmaceuticals), in Patients With Chronic Renal Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório Químico Farmacêutico Bergamo Ltda. (Industry)
Collaborators: Azidus Brasil (Industry)
Responsible Party: Marcelo A. C. Orlandi, Instituto de Nefrologia de Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEPBER0211
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Renal Failure
Keywords: heparin; renal insufficiency, chronic; extracorporeal dialysis; fibrinolytic agents; anticoagulants; aPTT
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Heparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actparin® - Laboratorio Bergamo (Experimental)
  Interventions: Biological: heparin sodium
- Heparin sodium - APP Pharmaceuticals (Active Comparator)
  Interventions: Biological: heparin sodium

INTERVENTIONS:
Biological: heparin sodium — 5000 UI/mL
  Arms: Actparin® - Laboratorio Bergamo
Biological: heparin sodium — 5000 UI/mL
  Arms: Heparin sodium - APP Pharmaceuticals

SUMMARY:
The purpose of this study is to investigate clinical non-inferiority, pharmacodynamic effect and safety of Actparin® (heparin sodium - Laboratório Químico Farmacêutico Bergamo Ltd.) compared to Heparin Sodium (APP Pharmaceuticals) in patients with renal failure under hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients research that agree to participate in the study and sign the informed consent form;
* Patients aged over 18 years, both sexes, regardless of color or social class;
* Patients with impaired renal function in chronic hemodialysis schedule of at least 3 times a week and giving the use of heparin in the prophylaxis of thrombosis in the system;
* Patients with laboratory results within specified acceptance criteria.

Exclusion Criteria:

* Patients who are taking part or took part in another clinical investigational study within 12 months;
* Hypersensitivity to heparin sodium and/or benzyl alcohol;
* History of active hemorrhage with alteration of blood coagulation, such as genetic disorders of coagulation system;
* History of disease that could aggravate or terminate the clinical manifestations, such as active peptic or gastric ulcer;
* Severe liver disease;
* Patients in cancer treatment;
* Pregnant and lactating women;
* Use of glucocorticoids over physiological dose;
* Use of other anticoagulants;
* Patients undergoing any surgery performed less than 15 days;
* History of non response or exacerbated response to heparin sodium;
* Patients who do not adapt to 150 UI/kg dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness in prevention of clotting in the extracorporeal circuit during hemodialysis | 4 weeks (12 consecutive sessions)

SECONDARY OUTCOMES:
Pharmacodynamic activity of heparin observed through aPTT marker | 4 weeks (sessions 1, 6 and 12)
Safety in use of heparin by monitoring adverse events | 5 weeks (12 consecutive sessions + 1 post treatment session)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A. C. Orlandi, Dr., Principal Investigator — Instituto de Nefrologia de Campinas
Locations (1):
- Instituto de Nefrologia de Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Blood thinners — http://www.nlm.nih.gov/medlineplus/bloodthinners.html
- See also: Dialysis — http://www.nlm.nih.gov/medlineplus/dialysis.html
- See also: Kidney failure — http://www.nlm.nih.gov/medlineplus/kidneyfailure.html
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Heparin — http://druginfo.nlm.nih.gov/drugportal/dpdirect.jsp?name=Heparin
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks